CLINICAL TRIAL: NCT04811352
Title: Readiness for a Pandemic, and Factors Associated With Substance Abuse During the COVID-19 Pandemic - A Cross-Sectional Study
Brief Title: Drug Abuse During the COVID-19 Pandemic.
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Uso_drogas
Record Dates: First submitted 2021-03-22; First posted 2021-03-23 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Substance Abuse; Stress, Psychological
Keywords: substance abuse; COVID-19; stress; economical impact
MeSH Terms: conditions — Substance-Related Disorders; Stress, Psychological; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pandemic we live through has put various sectors of the medical system and its tributaries to the test. The accumulation of external and internal stress has been completely correlated with the predisposition to psycho-emotional problems and, in turn, to drug use as an immature response for ego protection. That is why the economic, social, and psychological evaluation can help understand the current situation about drug abuse and how to help patients afflicted by it. The added stress of personal problems, work alterations, daily life in a pandemic, economic and varied responsibilities, and the understanding of the pandemic have predisposed and amplified the use of drugs to reduce emotional distress perceived by individuals. The hypothesis of this study is that the increment of stress and a lack of preparation for the pandemic are associated with increased drug abuse.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Willing to participate in the study
* Patient currently with a paying job

Exclusion Criteria:

* Patients without a paying job

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Mexican general population during the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Behaviour on drug and substance abuse | Baseline
  The survey inquires about the frequency and dosage of numerous substances such as coffee, alcohol, tobacco, and heroin since the pandemic started.
PHQ-9 Score | Baseline
  This inventory will be used to identify the presence and intensity of depressive disorders. The minimum score is 0, and the maximum score is 27.
GAD-7 Score | Baseline
  This questionnaire will be used to evaluate the presence and intensity of anxiety disorders. The minimum score is 0, and the maximum score is 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico